CLINICAL TRIAL: NCT00618280
Title: Social Cognition,Attentional Network and Nicotine Drug Dependency - A Pharmacological Clinical Trail
Acronym: NIKOGEN
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: NIKOGEN_HHU_2006
Record Dates: First submitted 2008-02-08; First posted 2008-02-20 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-03

CONDITIONS: Tobacco Use Disorder; Schizophrenia
MeSH Terms: conditions — Tobacco Use Disorder; Schizophrenia | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): schizophrenic and non schizophrenic patient stratified by smoking and non smoking will get nicotine and placebo on first day on the second day placebo and nicotine
  Interventions: Drug: nicotine nasal spray
- 2 (Placebo Comparator): schizophrenic and non schizophrenic patient stratified by smoking and non smoking will get nicotine and placebo on first day on the second day placebo and nicotine
  Interventions: Drug: nicotine nasal spray

INTERVENTIONS:
Drug: nicotine nasal spray — 0,5 mg nicotine nasal spray or placebo (pepperspray)
  Other Names: nicorette nasal spray

SUMMARY:
In the present study, we investigate healthy subjects and schizophrenic patients who frequently show very low attentional capacity with functional magnetic resonance imaging (fMRI) and electrophysiology (EEG) during attention-requiring tasks to assess the level of attentional network activity.

DETAILED DESCRIPTION:
Nicotine is improving attentional capacity which goes along with an activation of the attentional network in the brain. So far, however, it is unresolved whether nicotine is used for the purpose of self-medication by those nicotine-dependent subjects who suffer from subclinical or clinical attentional deficits which may sustain nicotine addiction. In the present study, we investigate healthy subjects and schizophrenic patients who frequently show very low attentional capacity with functional magnetic resonance imaging (fMRI) and electrophysiology (EEG) during attention-requiring tasks to assess the level of attentional network activity. It is anticipated that low attentional network activity (during baseline condition, after nicotine challenge and after withdrawal) predicts the degree of nicotine dependence including the strength of withdrawal symptoms and relapse rate after smoking cessation. In addition, we expect that functional variations within alpha4beta2 nAch receptor genotype are associated with attentional capacity and -by extension - with nicotine dependence.

Additionally Self-medication of attentional deficits and of increased stress vulnerability may contribute to nicotine-dependence both in schizophrenia patients and healthy subjects. However, very little is known about the effect of nicotine on stress in schizophrenia. In particular social stressors are highly relevant in schizophrenia often resulting in social withdrawal. A factor contributing to the stress-eliciting nature of social interaction is the misidentification of social information during communication with others. The present project aims at an investigation of nicotine effects on such social information processing and its neurophysiological correlates and on social stress responses. Using a 2x2-factorial design effects of nicotine vs. placebo are experimentally investigated in smoking schizophrenia patients in comparison to smoking healthy controls each after an overnight smoking deprivation. Nicotine will be administered by nasal spray delivering a systemic does of 2 mg nicotine. Event-related EEG potentials will be recorded during the presentation of pictures of facial affect and neutral control stimuli to assess social information processing and its neurophysiological correlates. In addition a videotaped semi-standardized conversation skills role-play test will be used as a social stress situation to assess self-reported and non-verbal affective responses.

ELIGIBILITY:
Inclusion Criteria:

* age 18-55
* informed consent
* negative drug-screening (cannabis, amphetamine, opiate, cocaine)
* no drug abuse in medical history for last 6 month
* no participation of subjects in other pharmacological trials within 6 weeks
* negative pregnancy test
* use of effective contraception within participation of trial
* normotonia (heart rate, RR)
* nicotine dependence (Fagerström >4)or not more than 20 cigarettes /lifetime
* nicotine (smoker serum > 2ng/mL)
* DSM-IV criteria for schizophrenia
* healthy subjects

Exclusion Criteria:

* known hypersensitivity towards nicotine or any substance of placebo preparation
* adenoids
* Rhinitis vaso.
* hypersensitivity of air passages
* cardiovascular diseases (defined)
* neurological diseases (defined)
* diabetes mellitus
* hyperthyreosis
* phaeochromocytoma
* Clozapine (schizophrenic)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2008-01; Primary Completion 2010-06 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Effect of nicotine or placebo in healthy subjects and schizophrenic patients on attentional network activity in brain with functional magnetic resonance imaging and EEG | after last subject out

SECONDARY OUTCOMES:
-Effect of nicotine on a4b2 nAch receptor genotype -Gene Expression of a4b2 nAch -effect of 24 h nicotine withdrawal on modulation special hormones -effect of nicotine on neurophysiological correlates of social stress | after last subject out

CONTACTS AND LOCATIONS:
Overall Officials: G. Winterer, Prof. Dr., Principal Investigator — Department of Psychiatry and Psychotherapy
Locations (2):
- Germany (2):
  - Psychiatrische Klinik und Poliklinik der Heinrich-Heine-Universität, Düsseldorf, North Rhine-Westphalia
  - Forschungszentrum Jülich GmbH, Jülich, North Rhine-Westphalia

REFERENCES:
- [Derived] Warbrick T, Mobascher A, Brinkmeyer J, Musso F, Stoecker T, Shah NJ, Fink GR, Winterer G. Nicotine effects on brain function during a visual oddball task: a comparison between conventional and EEG-informed fMRI analysis. J Cogn Neurosci. 2012 Aug;24(8):1682-94. doi: 10.1162/jocn_a_00236. Epub 2012 Mar 27. PMID 22452559
- [Derived] Luckhaus C, Henning U, Ferrea S, Musso F, Mobascher A, Winterer G. Nicotinic acetylcholine receptor expression on B-lymphoblasts of healthy versus schizophrenic subjects stratified for smoking: [3H]-nicotine binding is decreased in schizophrenia and correlates with negative symptoms. J Neural Transm (Vienna). 2012 May;119(5):587-95. doi: 10.1007/s00702-011-0743-1. Epub 2011 Dec 11. PMID 22160487
- See also: Related Info — http://www.nicotine-research.com